CLINICAL TRIAL: NCT01643954
Title: Retrospective/Prospective Analysis of Surgical Outcomes of Robotic Prostatectomy at Ohio State University/The James.
Brief Title: Retrospective/Prospective Analysis of Surgical Outcomes of Robotic Prostatectomy at The James
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Steven Clinton, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OSU-08108
Record Dates: First submitted 2012-05-08; First posted 2012-07-18 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-12

CONDITIONS: Prostate Cancer
Keywords: prostatectomy; surgery; prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Laparoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (No Intervention): Patients with prostate cancer who have undergone robotic radical prostatectomy at The Arthur G. James Cancer Hospital and Solove Research Institute, The Ohio State University Medical Center.
- Arm B (Other): Patients with prostate cancer that will undergo robotic radical prostatectomy at The Arthur G. James Cancer Hospital and Solove Research Institute, The Ohio State University Medical Center .
  Interventions: Procedure: robotic radical prostatectomy

INTERVENTIONS:
Procedure: robotic radical prostatectomy — robotic assisted surgery
  Other Names: laparoscopic surgery; The da Vinci system
  Arms: Arm B

SUMMARY:
This is a retrospective/prospective Analysis of surgical outcomes of robotic prostatectomy.

DETAILED DESCRIPTION:
This retrospective / prospective study will allow us to collect and analyze the presurgical, peri-operative, and outcome data of patients who undergo robotic radical prostatectomy at The Arthur G. James Cancer Hospital and Solove Research Institute, The Ohio State University Medical Center, beginning February 2008 onwards.

ELIGIBILITY:
ARM A:

Inclusion Criteria:

* Patients with prostate cancer who have undergone robotic radical prostatectomy at The Arthur G. James Cancer Hospital and Solove Research Institute, The Ohio State University Medical Center.
* Ability to understand and willingness to sign the written informed consent document.
* 18 years and older

ARM B:

Inclusion Criteria:

* Patients with prostate cancer that will undergo robotic radical prostatectomy at The Arthur G. James Cancer Hospital and Solove Research Institute, The Ohio State University Medical Center.
* Ability to understand and willingness to sign the written informed consent document.
* 18 years and older

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1531 (Estimated)
Dates: Start 2008-09-23 (Actual); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Collect and analyze descriptive characteristics of patient population and summarize patient outcome data. | up to 20 years

SECONDARY OUTCOMES:
Correlate the patient characteristics to the surgical outcomes. | up to 20 years
Determine the overall survival | up to 20 years
Determine the rate of local recurrence in patients undergoing robotic prostatectomy and compare these metrics to historical controls. | up to 20 years
disease- free survival | up to 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Clinton, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

REFERENCES:
- See also: Jamesline — http://cancer.osu.edu